CLINICAL TRIAL: NCT00096291
Title: Neoadjuvant Chemotherapy in Palpable Breast Cancer: Evaluation of Physiologic, Radiologic, and Molecular Markers in Predicting Response
Brief Title: Neoadjuvant Chemotherapy Using Doxorubicin and Paclitaxel in Treating Women With Large Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Alphonse Taghian, MD, PhD, Principle Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CDR0000382123; P50CA089393 (NIH); P30CA006516 (NIH); DFCI-99278
Record Dates: First submitted 2004-11-09; First posted 2004-11-09 (Estimated); Last update posted 2017-04-10 (Actual); Status verified 2017-04

CONDITIONS: Breast Cancer
Keywords: stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sequence Doxorubicin followed by Paclitaxel (Active Comparator): Patients will be randomized into 2 groups based on sequence of neoadjuvant chemotherapy:
  Doxorubicin followed by Paclitaxel versus Paclitaxel followed by Doxorubicin
  Interventions: Other: Doxorubicin followed by Paclitaxel; Other: Paclitaxel followed by Doxorubicin
- Sequence of neoadjuvant CT: Paclitaxel followed by Doxorubicin (Other): Patients will be randomized into 2 groups based on sequence of neoadjuvant chemotherapy:
  Doxorubicin followed by Paclitaxel versus Paclitaxel followed by Doxorubicin
  Interventions: Other: Paclitaxel followed by Doxorubicin

INTERVENTIONS:
Other: Doxorubicin followed by Paclitaxel — Patients will be randomized into 2 groups based on sequence of neoadjuvant chemotherapy:
  Doxorubicin followed by Paclitaxel Paclitaxel followed by Doxorubicin
  Arms: Sequence Doxorubicin followed by Paclitaxel
Other: Paclitaxel followed by Doxorubicin — Patients will be randomized into 2 groups based on sequence of neoadjuvant chemotherapy:
  Doxorubicin followed by Paclitaxel versus Paclitaxel followed by Doxorubicin

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as doxorubicin and paclitaxel, work in different ways to stop tumor cells from dividing so they stop growing or die. Giving chemotherapy before and after surgery may shrink the tumor so it can be removed and may kill any tumor cells remaining after surgery.

PURPOSE: This randomized phase II trial is comparing two different regimens of doxorubicin and paclitaxel to see how well they work in treating women who are undergoing surgery for breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine whether tumors in women with palpable invasive breast cancer with wild type p53 are more sensitive to doxorubicin than to paclitaxel when given as sequential single-agent neoadjuvant chemotherapy.
* Determine whether tumors with inactivated p53 are more sensitive to paclitaxel than to doxorubicin when given as sequential single-agent neoadjuvant chemotherapy in these patients.

Secondary

* Correlate other biological markers (physiological and molecular) with tumor response in patients treated with these regimens.
* Determine changes in these biological markers during and after neoadjuvant chemotherapy in these patients.
* Compare breast MRI, in terms of assessing tumor response, with physical exam, mammogram, and ultrasound in patients treated with these regimens.
* Determine whether there are MRI indicators (e.g., tumor morphology or lesion enhancement) that are predictive of response in patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to tumor size (> 5 cm vs ≤ 3-5 cm) and presence of palpable regional lymph nodes (yes vs no). Patients are randomized to 1 of 2 treatment arms.

All patients undergo biopsy, bilateral mammogram, MRI, ultrasound, blood marker, molecular (gene microarrays and functional p53 status), and physiologic studies before initiation of neoadjuvant chemotherapy. Some of these studies are repeated after completion of treatment with the first chemotherapeutic agent and after completion of treatment with the second chemotherapeutic agent as outlined below.

* Arm I: Patients receive doxorubicin IV on days 1, 15, 29, and 43. Patients with no residual tumor (indicated by clinical evaluation and radiologic studies) after completion of doxorubicin undergo definitive surgery. After surgery, patients receive paclitaxel IV over 1 hour on days 1, 8, 15, 22, 29, 36, 43, 50, and 57.

Patients with residual tumor > 2 cm after completion of doxorubicin undergo 8-12 core needle biopsies. Patients with residual tumor < 2 cm after completion of doxorubicin undergo 4-6 core needle biopsies. After core needle biopsies, patients receive paclitaxel as above.

* Arm II: Patients receive paclitaxel IV over 1 hour on days 1, 8, 15, 22, 29, 36, 43, 50, and 57. Patients with no residual tumor (indicated by clinical evaluation and radiologic studies) after completion of paclitaxel undergo definitive surgery. After surgery, patients receive doxorubicin IV on days 1, 15, 29, and 43.

Patients with residual tumor > 2 cm after completion of paclitaxel undergo 8-12 core needle biopsies. Patients with residual tumor < 2 cm after completion of paclitaxel undergo 4-6 core needle biopsies. After core needle biopsies, patients receive doxorubicin as above.

In both arms, treatment continues in the absence of disease progression or unacceptable toxicity.

Samples from core needle biopsies are analyzed by microarray analysis for gene expression profiles.

Patients are followed every 6 months for 5 years.

PROJECTED ACCRUAL: A total of 100 patients (50 per treatment arm) will be accrued for this study within 4-5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of invasive breast cancer

  * Tumor ≥ 3 cm and palpable

    * Multiple masses are allowed provided at least 1 mass is ≥ 3 cm
  * Clinically positive axillary or supraclavicular lymph nodes allowed
  * Fine needle aspiration or core needle biopsy positive for invasive breast cancer AND/OR fine needle aspiration of lymph nodes positive
* HER2/neu-positive OR negative
* No inflammatory breast cancer
* No distant metastases
* Hormone receptor status:

  * Estrogen receptor (ER)-positive OR ER-negative

PATIENT CHARACTERISTICS:

Age

* 18 and over

Sex

* Female

Menopausal status

* Premenopausal or postmenopausal

Performance status

* Karnofsky 60-100%

Life expectancy

* Not specified

Hematopoietic

* Granulocyte count ≥ 1,000/mm^3
* Platelet count ≥ 100,000/mm^3

Hepatic

* Bilirubin ≤ 2 times upper limit of normal (ULN)
* SGOT ≤ 2 times ULN

Renal

* Not specified

Cardiovascular

* LVEF ≥ 50%
* No congestive heart failure
* No serious conduction system abnormality
* No other significant cardiovascular disease

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Patients with other prior or concurrent malignancies allowed provided they have received no prior chemotherapy AND they are likely to have been cured from a prior malignancy
* No severe medical or psychiatric condition that would preclude study compliance
* No known HIV positivity

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior chemotherapy

Endocrine therapy

* No prior hormonal therapy for breast cancer

Radiotherapy

* No prior radiotherapy for this malignancy

Surgery

* Not specified

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2000-02; Primary Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
•Determine whether tumors in women with palpable invasive breast cancer with wild type p53 are more sensitive to doxorubicin than to paclitaxel when given as sequential single-agent neoadjuvant chemotherapy | asses pathological response to neoadjuvant chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Alphonse G. Taghian, MD, PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts

REFERENCES:
- [Result] Taghian AG, Abi-Raad R, Assaad SI, Casty A, Ancukiewicz M, Yeh E, Molokhia P, Attia K, Sullivan T, Kuter I, Boucher Y, Powell SN. Paclitaxel decreases the interstitial fluid pressure and improves oxygenation in breast cancers in patients treated with neoadjuvant chemotherapy: clinical implications. J Clin Oncol. 2005 Mar 20;23(9):1951-61. doi: 10.1200/JCO.2005.08.119. PMID 15774788
- [Result] Yeh E, Slanetz P, Kopans DB, Rafferty E, Georgian-Smith D, Moy L, Halpern E, Moore R, Kuter I, Taghian A. Prospective comparison of mammography, sonography, and MRI in patients undergoing neoadjuvant chemotherapy for palpable breast cancer. AJR Am J Roentgenol. 2005 Mar;184(3):868-77. doi: 10.2214/ajr.184.3.01840868. PMID 15728611